CLINICAL TRIAL: NCT01131806
Title: Comparing Treatment Efficacy With High and Medium Dose of Fluticasone in Combination With Salmeterol in COPD Patients
Brief Title: Comparing Treatment Efficacy With HD/MD Flu Plus Sal in Chronic Obstructive Pulmonary Disease (COPD) Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Collaborators: National Taiwan University Hospital (Other); Far Eastern Memorial Hospital (Other)
Responsible Party: Diahn-Warng PERNG/ Chief, Division of Respiratory Care Unit, Veterans General Hospital-TAIPEI, Department of Chest
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VGHIRB No. 98-10-16; CM981016 (Other: Veterans General Hospital-TAIPEI)
Record Dates: First submitted 2010-05-25; First posted 2010-05-27 (Estimated); Last update posted 2010-07-08 (Estimated); Status verified 2010-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: chronic obstructive pulmonary disease; lung function change FEV1 FVC; acute exacerbation; life quality questionnaire
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Fluticasone; Salmeterol Xinafoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MD Flu/Sal (Active Comparator): fluticasone125 mcg/ salmeterol 25 mcg 2puffs (medium dose group) inhaled twice daily; salbutamol evohaler allowed from 100 to 400 mcg for inhalation as needed basis.
  Interventions: Drug: fluticasone/ salmeterol 125/25 mcg/puff
- HD Flu/Sal (Experimental): fluticasone 250 mcg/salmeterol 25 mcg 2puffs (high dose group) inhaled twice daily; salbutamol evohaler allowed from 100 to 400 mcg for inhalation as needed basis.
  Interventions: Drug: fluticasone/ salmeterol 250/25 mcg/puff

INTERVENTIONS:
Drug: fluticasone/ salmeterol 125/25 mcg/puff — fluticasone 125mcg/salmeterol 25mcg 2puffs/day x 52 weeks
  Other Names: Seretide evohaler 125(GlaxoSmithKline)
  Arms: MD Flu/Sal
Drug: fluticasone/ salmeterol 250/25 mcg/puff — fluticasone 250mcg/salmeterol 25mcg 2puffs/day x 52 weeks
  Other Names: Seretide evohaler 250(GlaxoSmithKline)
  Arms: HD Flu/Sal

SUMMARY:
Chronic obstructive pulmonary disease is characterized as inflammatory airway with not fully reversible airflow limitation.Combination treatment with inhaled corticosteroid (ICS) and long-acting β2 agonists (LABA)attains an improved control of symptoms and lung function, that are superior to those associated with either drug alone. However, the treatment efficacy between high and medium dose of inhaled corticosteroid in combination of LABA is still unknown. The aim of the current study is to investigate the treatment efficacy with high and medium dose of fluticasone in combination with salmeterol in COPD patients.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a major cause of morbidity and the use of health care resources worldwide. It is characterized by chronic progressive symptoms, airflow obstruction, and impaired health status, which is worse in those who have frequent, acute episodes of symptom exacerbation. Treatment for COPD is focused on minimizing risk factors, improving symptoms, and preventing exacerbations.

Pulmonary inflammation is the key factor in COPD. Inhaled long-acting β2 agonists (LABA) improve airflow obstruction, control of symptoms, and health status in patients with COPD over 3 to 4 months. Inhaled corticosteroids (ICS) are currently the most popular anti-inflammatory medications for use in symptomatic patients with COPD. Previous large scaled randomized control study discovered long-term use of ICS didn't modified annual decline of lung function in COPD patients, but may reduce the frequency of exacerbations, especially when combined with an LABA.

Combination treatment with ICS and LABA has been widely used for patients with COPD and attains an improved control of symptoms and lung function, with no greater risk of side-effects than that of treatment with either component alone. Combined ICS/LABA will result in better treatment effects that are superior to those associated with either drug alone. However, the treatment efficacy between high and medium dose of inhaled corticosteroid in combination of LABA is still unknown. The aim of the current study is to investigate the treatment efficacy with high and medium dose of fluticasone in combination with salmeterol in COPD patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients aged ≧ 40 years.
* Current or ex-smoker, with smoking history ≧ 10 pack- years
* COPD (FEV1/FVC < 70%) patients with post-bronchodilator FEV1 ≦ 70% predicted value, without bronchial reversibility (≦10% increase post bronchodilator).

Exclusion Criteria:

* Diagnosis or suspicion of sleep apnea
* Concurrent rhinitis, eczema, and asthma
* Clinically overt bronchiectasis, lung cancer, active tuberculosis, or other known specific pulmonary disease
* A chest X-ray indicating diagnosis other than COPD that might interfere with the study.
* Major disease abnormalities are uncontrolled on therapy.
* Alcohol or medication abuse.
* Patients had lower respiratory tract infections or received systemic steroid in the 4 weeks prior to the commencement of study.
* Unable or unwilling to comply with all protocol specified procedures.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2009-12; Primary Completion 2010-11 (Estimated); Study Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
The change of lung function parameters(FEV1&FVC) at different time points | baseline, week 12, 28 and 52
  The changes of lung function parameters, including post bronchodilation forced expiratory volume in first second (FEV1) and forced vital capacity (FVC), at different time points, including baseline, 12th week, 28th week, and ending (52th week).

SECONDARY OUTCOMES:
Annual rate of acute exacerbations | 1 year
  total numbers of acute exacerbation throughout the study year
Life quality evaluation | baseline, week 12, 28, and 52
  The changes of Health-related quality of life assessed by CAT questionnaire before and after treatment.
Annual incidence of community-acquired pneumonia | 1 year
  Annual incidence of community-acquired pneumonia throughout the study year

CONTACTS AND LOCATIONS:
Overall Officials: Diahn-Warng Perng, PhD, Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Chest department, Veteran General Hospital-TAIPEI, Taipei, Taiwan, Taiwan

REFERENCES:
- [Background] Calverley PM, Anderson JA, Celli B, Ferguson GT, Jenkins C, Jones PW, Yates JC, Vestbo J; TORCH investigators. Salmeterol and fluticasone propionate and survival in chronic obstructive pulmonary disease. N Engl J Med. 2007 Feb 22;356(8):775-89. doi: 10.1056/NEJMoa063070. PMID 17314337
- [Background] Keating GM, McCormack PL. Salmeterol/fluticasone propionate: a review of its use in the treatment of chronic obstructive pulmonary disease. Drugs. 2007;67(16):2383-405. doi: 10.2165/00003495-200767160-00006. PMID 17983257
- [Background] Hanania NA, Darken P, Horstman D, Reisner C, Lee B, Davis S, Shah T. The efficacy and safety of fluticasone propionate (250 microg)/salmeterol (50 microg) combined in the Diskus inhaler for the treatment of COPD. Chest. 2003 Sep;124(3):834-43. doi: 10.1378/chest.124.3.834. PMID 12970006
- [Background] Szafranski W, Cukier A, Ramirez A, Menga G, Sansores R, Nahabedian S, Peterson S, Olsson H. Efficacy and safety of budesonide/formoterol in the management of chronic obstructive pulmonary disease. Eur Respir J. 2003 Jan;21(1):74-81. doi: 10.1183/09031936.03.00031402. PMID 12570112